CLINICAL TRIAL: NCT04080947
Title: The Leukotriene Receptor Antagonist Montelukast in the Treatment of Non-alcoholic Steatohepatitis: A Proof-of-Concept, Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: The Leukotriene Receptor Antagonist Montelukast in the Treatment of Non-alcoholic Steatohepatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sadat City University (Other)
Responsible Party: Principal Investigator, Mahmoud Samy Abdallah, Lecturer of Clinical Pharmacy, PhD., Sadat City University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 002017
Record Dates: First submitted 2019-08-31; First posted 2019-09-06 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Steatohepatitis, Nonalcoholic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): 26 patients will receive placebo (Control group)
  Interventions: Drug: Control group
- Montelukast group (Experimental): 26 patients will receive montelukast 10 mg/ day
  Interventions: Drug: Montelukast group

INTERVENTIONS:
Drug: Control group — patients received matching-image placebo once daily at bedtime for 12 weeks.
  Arms: Control group
Drug: Montelukast group — patients received montelukast (10-mg chewable tablet) once daily at bedtime for 12 weeks.
  Arms: Montelukast group

SUMMARY:
The aim of the current study is to evaluate the safety and efficay of Montelukast in treatment of patients with fatty liver disease.

ELIGIBILITY:
Inclusion Criteria:

- The inclusion criteria were adult patients (age >18 years old) of both sexes, overweight/obese subjects with presence of evidence of hepatic steatosis by imaging (increased liver echogenicity, stronger echoes in the hepatic parenchyma, vessel blurring, and narrowing of the lumen of the hepatic veins). Patients with mild to moderate elevation in aminotransferase activities (> 2 but <5 times upper limit of normal), hepatic steatosis index (HIS) >36, Fibro-scan score >7 kpa and <12.5 kpa (F0-F3), and HAIR score of 2 or 3 were included in the study.

Exclusion Criteria:

- The exclusion criteria included smokers, patients with secondary hepatic fat accumulation which results from using steatogenic medications or hereditary disorders. Alcohol consumers, patients with Wilson's disease, hemochromatosis, viral hepatitis, decompensated liver disease, inflammatory diseases, diabetes, depression and patients with other comorbid conditions that elevate transaminases (congestive heart failure and malignancy) pregnancy and lactating women were excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Fibro-scan score | At baseline and after 12 weeks of intervention
  change in liver stiffness measurement (Fibro-scan score)
Liver Panel | after 12 weeks of intervention
  Alanine aminotransferase (ALT) and Aspartate Aminotransferase (AST) will be evaluated in U/L

SECONDARY OUTCOMES:
HOMA-IR | after 12 weeks of intervention
  Homeostatic Model Assessment of Insulin Resistance
8-OHdG | after 12 weeks of intervention
  Serum level of 8-OHdG
TNF-Alpha | after 12 weeks of intervention
  Serum level of TNF-Alpha
hyaluronic acid | after 12 weeks of intervention
  Serum level of hyaluronic acid
TGF-β1 | after 12 weeks of intervention
  Serum level of TGF-β1
Assessment of drugs tolerability: Side effects | after 12 weeks of intervention
  Side effects of montelukast

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Derived] Abdallah MS, Eldeen AH, Tantawy SS, Mostafa TM. The leukotriene receptor antagonist montelukast in the treatment of non-alcoholic steatohepatitis: A proof-of-concept, randomized, double-blind, placebo-controlled trial. Eur J Pharmacol. 2021 Sep 5;906:174295. doi: 10.1016/j.ejphar.2021.174295. Epub 2021 Jun 30. PMID 34214585